CLINICAL TRIAL: NCT04173000
Title: Web Based Tools to Improve Medication Continuity in Adolescents With ADHD
Brief Title: Tools to Improve Medication Continuity in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-0172
Record Dates: First submitted 2019-11-05; First posted 2019-11-21 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open Label Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All adolescent/parent dyads enrolled at each practice will have access to the meHealth for ADHD software without medication continuity tools prior to being given access to the medication continuity tools.
  Interventions: Other: Mehealth for ADHD software with medication continuity tools; Other: Mehealth for ADHD software without medication continuity tools

INTERVENTIONS:
Other: Mehealth for ADHD software with medication continuity tools — Medication continuity tools integrated within the mehealth for ADHD software will assess factors influencing medication continuity for each adolescent and recommends tools to address relevant factors. Tools include 1) a system to track outcomes and resolve uncertainty about the need for and/or benefit from medicine, 2) a module to address stigma, 3) a module to help manage side effects, and 4) reminders to take medicine and/or request refills.
Other: Mehealth for ADHD software without medication continuity tools — The mehealth for ADHD software has multiple functionalities including 1) online training regarding the American Academy of Pediatrics (AAP) ADHD guidelines; 2) an ADHD workflow wizard that guides pediatricians through the creation of an efficient office workflow to deliver quality ADHD care; 3) online collection of parent- and teacher-report ADHD rating scales for the assessment of ADHD as well as monitoring response to medication treatment; 4) integrated algorithms that automatically score rating scales in real time and provide pediatricians with assessment and treatment reports as well as immediate warnings; 5) a communication feature that allows parents, teachers, and pediatricians to communicate with each other; 6) an online pediatrician "report card"; and 7) a Plan-Do-Study-Act wizard that allows pediatricians to select a practice behavior to improve based on their report card and guides them through the creation of small tests of change to improve their office systems.

SUMMARY:
Medication is an efficacious treatment strategy for adolescents with attention-deficit/hyperactivity disorder (ADHD), however use significantly declines during adolescence when the consequences of ADHD are most severe (e.g. dropping out of school, delinquency, etc.). The Unified Theory of Behavior Change (UTBC) has been proposed as a conceptual model to explain the mechanism underlying ADHD medication adherence and to guide the development of interventions to improve the continuity of treatment. The UTBC is a well-established and empirically tested model that identifies factors that influence an individual's intention to perform a behavior as well as factors that influence whether a behavior is actually carried out. Indeed, the research team's preliminary data support the relevance of pre-intention factors and implementation factors for medication continuity among adolescents with ADHD. Currently, no evidence-based interventions target medication continuity for adolescents with ADHD. The objective of this study is to test a multi-component intervention that systematically identifies and targets aspects of the UTBC model most relevant for each adolescent with poor ADHD medication continuity. The central hypothesis is that the tailored intervention will support ADHD medication continuity. The study will conduct an open label trial among adolescents with poor medication continuity to test whether the intervention engages the mechanism underlying medication continuity and improves outcomes.

ELIGIBILITY:
Inclusion Criteria:

* First prescribed ADHD medicine more than one year prior to enrollment
* Registered on myADHDportal.com at practice participating in study
* Filled at least one prescription for a stimulant medication in the past year

Exclusion Criteria:

* More than 80% of days covered with medicine over past one year
* Poor understanding level: The participant and parent cannot understand or follow instructions given in the study.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: All parent/adolescent dyads enrolled at each practice will have access to the meHealth for ADHD software without medication continuity tools prior to being given access to the medication continuity tools.
  Mehealth for ADHD software with medication continuity tools: Medication continuity tools integrated within the mehealth for ADHD software will assess factors influencing medication continuity for each adolescent and recommends tools to address relevant factors. Tools include 1) a system to track outcomes and resolve uncertainty about the need for and/or benefit from medicine, 2) a module to address stigma, 3) a module to help manage side effects, and 4) reminders to take medicine and/or request refills.
Period: Overall Study
Arm/Group | Intervention
Started | 8 (8 adolescent-parent dyads with a total of 16 participants)
Completed | 8 (8 adolescent-parent dyads with a total of 16 participants)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 8 adolescent-parent dyads included a total of 16 participants
Arm/Group | Intervention
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years]
  Adolescent | 13.60 (1.70)
  Parent | 44.62 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Adolescent: Female | 3
  Adolescent: Male | 5
  Parent: Female | 8
  Parent: Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: Hispanic or Latino | 0
  Adolescent: Not Hispanic or Latino | 8
  Adolescent: Unknown or Not Reported | 0
  Parent: Hispanic or Latino | 0
  Parent: Not Hispanic or Latino | 8
  Parent: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Adolescent: American Indian or Alaska Native | 0
  Adolescent: Asian | 0
  Adolescent: Native Hawaiian or Other Pacific Islander | 0
  Adolescent: Black or African American | 0
  Adolescent: White | 5
  Adolescent: More than one race | 3
  Adolescent: Unknown or Not Reported | 0
  Parent: American Indian or Alaska Native | 0
  Parent: Asian | 0
  Parent: Native Hawaiian or Other Pacific Islander | 0
  Parent: Black or African American | 1
  Parent: White | 7
  Parent: More than one race | 0
  Parent: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days Covered With Medicine
Description: This will be calculated based pharmacy dispensing records
Time Frame: An average of 4 months
Population: Missing data for 1 adolescent
Measure: Mean (Full Range); unit: Proportion of days covered with medicine
Arm/Group | Intervention
Number analyzed (Participants) | 7
Proportion of days covered with medicine | 0.69 [0.44 to 0.98]

2. Secondary Outcome: Fidelity to Intended Use of Intervention Components
Description: Proportion of intervention components completed relative to the components that were recommended by the portal based on adolescent/parent responses to the assessment battery.
Time Frame: An average of 4 months
Measure: Mean (Full Range); unit: Proportion of intervention components
Arm/Group | Intervention
Number analyzed (Participants) | 16
Proportion of intervention components | 0 [0 to 0]

3. Secondary Outcome: Change in Pre-intention Factors of Unified Theory of Behavior Change Influencing Medication Continuity
Description: Adolescent and parent self-report on a 1-5 or 1-7-point scale, depending on the item. Items were re-scaled to a 1 (signifying less belief) to 5 (signifying stronger belief) scale. Individual items measure specific attitudes, subjective norms, and perceived behavioral control. Items were coded so that higher scores aligned with increased perceived advantages of performing the behavior and behavioral control around taking ADHD medicine. We calculated the average score of the total items (Adolescent report = 19 items; Parent report = 17 items). Range of change score is (-4) to (+4).
Time Frame: At baseline and 4 months later
Population: Missing data for 1 parent/adolescent dyad and 1 adolescent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale
  Adolescent: number analyzed (Participants) | 6
  Adolescent | -0.19 (0.27)
  Parent: number analyzed (Participants) | 7
  Parent | -0.14 (0.37)

4. Secondary Outcome: Change in Intention to Take/Give ADHD Medicine Regularly
Description: Adolescent and parent self-report on a 1-7-point scale. Items were re-scaled to a 1 (signifying less intention) to 5 (signifying stronger intention) scale. Items were coded so that higher scores aligned with stronger intention to take ADHD medicine every school day, weekend day, and during school vacations. We calculated the average score of the 3 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and 4 months later
Population: Missing data for 1 parent/adolescent dyad and 1 adolescent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale
  Adolescent: number analyzed (Participants) | 6
  Adolescent | -0.07 (1.28)
  Parent: number analyzed (Participants) | 7
  Parent | 0.03 (0.55)

5. Secondary Outcome: Change in Adolescent Report of Medication Barriers
Description: Adolescent self-report on Adolescent Medication Barriers Scale using a 1-5-point Likert Scale. 1 indicates strong agreement and 5 indicates strong disagreement, with higher scores indicating less barriers. Items were coded so that higher scores aligned with increased organizational skills, salience of behavior, and routine around taking ADHD medicine. We calculated the average score of the 8 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and 4 months later
Population: Missing data for 2 adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 6
score on a scale | -0.44 (1.03)

6. Secondary Outcome: Change in Parent Report of Medication Barriers
Description: Parent self-report on Parent Medication Barriers Scale using a 1-5-point Likert Scale. 1 indicates strong agreement and 5 indicates strong disagreement, with higher scores indicating less barriers. Items were coded so that higher scores aligned with increased adolescent organizational skills, salience of behavior, and routine around taking ADHD medicine. We calculated the average score of the 9 items. Range of change score is (-4) to (+4).
Time Frame: At baseline and 4 months later
Population: Missing data for 1 parent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 7
score on a scale | 0.25 (0.51)

7. Secondary Outcome: Change in Medication Diversion
Description: Adolescent self-report of the number of occasions of giving away, trading, or selling ADHD medicine to someone for whom it was not prescribed.
Time Frame: At baseline and 4 months later
Population: Missing data for 2 adolescents
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Intervention
Number analyzed (Participants) | 6
Events | 0 (0)

8. Secondary Outcome: Change in Decision Making Involvement Scale
Description: Adolescent and Parent self-report. The scale contains the following subscales: "Child Seek" (e.g. child asks for an opinion or information from the parent), "Child Express" (e.g. child expresses an opinion or information to the parent), "Parent Seek" (e.g. parent asks for an opinion or information from child), "Parent Express" (e.g. parent expresses advice, an opinion, or information to the child), and "Joint/Options" (e.g. negotiation and brainstorming between child and parent). Each subscale produces a score which ranges from 1 to 4 with higher scores indicating more of that behavior.
Time Frame: At baseline and 4 months later
Population: Missing data for 1 parent/adolescent dyad and 1 adolescent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
score on a scale
  Adolescent: Child Seek: number analyzed (Participants) | 6
  Adolescent: Child Seek | -0.39 (0.49)
  Adolescent: Child Express: number analyzed (Participants) | 6
  Adolescent: Child Express | -0.22 (0.69)
  Adolescent: Parent Seek: number analyzed (Participants) | 6
  Adolescent: Parent Seek | -0.08 (0.68)
  Adolescent: Parent Express: number analyzed (Participants) | 6
  Adolescent: Parent Express | -0.23 (0.67)
  Adolescent: Joint/Options: number analyzed (Participants) | 6
  Adolescent: Joint/Options | 0.07 (0.86)
  Parent: Child Seek: number analyzed (Participants) | 7
  Parent: Child Seek | -0.19 (0.63)
  Parent: Child Express: number analyzed (Participants) | 7
  Parent: Child Express | 0 (1)
  Parent: Parent Seek: number analyzed (Participants) | 7
  Parent: Parent Seek | 0.18 (0.66)
  Parent: Parent Express: number analyzed (Participants) | 7
  Parent: Parent Express | 0.17 (0.58)
  Parent: Joint/Options: number analyzed (Participants) | 7
  Parent: Joint/Options | -0.23 (0.34)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT04173000/Prot_001.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04173000/SAP_002.pdf
  • Informed Consent Form (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT04173000/ICF_000.pdf